CLINICAL TRIAL: NCT03649347
Title: Bringing Exposure Therapy for Animal Phobias to Real-Life Context With Augmented Reality
Brief Title: Bringing Exposure Therapy to Real-Life Context With Augmented Reality
Acronym: ARET
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Data collection was completed for the spider arm of the study. No participants were recruited for snake phobia data collection due to the COVID-19 pandemic halting in-person research activities.
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Arash Javanbakht, Director of Stress, Trauma, and Anxiety Research Clinic, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1711000968
Record Dates: First submitted 2018-04-21; First posted 2018-08-28 (Actual); Results first posted 2022-03-07 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-03

CONDITIONS: Phobias Snakes; Phobias Spiders
Keywords: Exposure therapy; Technology; Telemedicine
MeSH Terms: conditions — Arachnophobia

STUDY DESIGN:
Intervention Model Description: 15 AR Therapy Intervention for Spider Phobia vs 15 No Treatment Control Group for Spider Phobia; 30 intervention vs 30 non intervention control group for fear of snakes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AR Therapy Intervention for Spider Phobia (Experimental): AR Therapy Intervention participants first complete a behavioral approach test (BAT). They approach a live spider to get as close as they comfortably can. This BAT provides a baseline measure of the degree of fear of spiders; the BAT is not a form of exposure therapy. Participants then complete exposure therapy using an augmented reality (AR) headset. A therapist controls the AR paradigm, placing virtual spiders in a participant's real environment as a method of exposure therapy. Once a participant's anxiety is reduced to low, stable levels (as measured by the participant's subjective units of distress assessed at intervals during session), the participant then completes a second BAT to measure their degree of fear immediately following AR therapy. The difference between the first and second BAT are used to assess the efficacy of the AR exposure therapy treatment. One month later, the AR Therapy Intervention participants complete a third BAT to assess for treatment efficacy over time.
  Interventions: Behavioral: Augmented reality exposure therapy
- No Treatment Control Group for Spider Phobia (No Intervention): The No Treatment Control group participants do not receive any AR exposure therapy for the duration of the study. These participants complete a behavioral approach test (BAT) at their first study visit, during which they approach a live spider as close as they comfortably can. This BAT provides a baseline measure of the degree of fear of spiders; the BAT is not a form of exposure therapy. One month later, the No Treatment Control group participants return for a second BAT to assess the degree to which their fear has changed as a function of time, in the context of NOT receiving any exposure therapy. After completion of the second BAT at this one-month follow-up visit, these participants are offered the opportunity for some form of exposure therapy following the conclusion of the study.
- AR Therapy Intervention for Snake Phobia (Experimental): Augmented reality (AR) exposure therapy involves placing virtual objects in the participant's real environment as a method of exposure therapy. The AR therapy intervention group will complete an exposure therapy session using an augmented reality headset. The participant will work with the therapist, who will control the augmented reality paradigm and cater the exposure to the needs of the participant. The exposure therapy session will be as long as needed to reduce anxiety to low and stable levels, as measured by the participant's subjective units of distress.
  Interventions: Behavioral: Augmented reality exposure therapy
- No Treatment Control Group for Snake Phobia (No Intervention): This will be a waitlist control group that will receive no treatment for the duration of the study, however they will be offered the opportunity for some form of exposure therapy following the conclusion of the study (1 month).

INTERVENTIONS:
Behavioral: Augmented reality exposure therapy — Exposure therapy via utilization of augmented reality. Virtual objects will be placed on the patient's real environment for exposure therapy.
  Arms: AR Therapy Intervention for Snake Phobia; AR Therapy Intervention for Spider Phobia

SUMMARY:
In this patented project, U.S. Patent No. 10,839,707, the investigators will develop an augmented reality exposure therapy method for arachnophobia, and fear of snakes, to test in the clinic. The platform will include a software that allows the clinician (psychiatrist/therapist) to position virtual objects in the real environment of the patient with the above mentioned phobias while the patient is wearing the augmented reality (AR) device. Then the clinician will lead the patient through steps of exposure therapy to the fear objects. The investigators will then measure the impact of treatment and compare to before treatment measures of fear of the phobic object.

Exposure therapy is the most evidence-based treatment for specific phobias, social phobia, obsessive-compulsive disorder (OCD), and posttraumatic stress disorder (PTSD). The core principle is patient's exposure to the feared objects/situations guided by a clinician. For example, in arachnophobia, patient is exposed to pictures of spiders printed or on a computer screen- or if available, view of a real tarantula in the office. Gradually, patient tolerates viewing/approaching the spider from a closer distance, and fear response extinguishes. The clinician has a crucial role in signaling safety to the patient, as well as providing support and coaching. This treatment is limited by multiple factors: 1) limited access to feared objects/situations in the clinic, 2) even when feared objects are available, they are not diverse (e.g. different types and colors of spiders), which limits generalization of safety learning, 3) when available, clinician has very limited control over behaviors of the feared objects (e.g. spider/snake), 4) safety learning is limited to the clinic office context, and contextualization of safety learning to real life experiences is left to the patient to do alone, which often does not happen. This is specifically important in conditions such as PTSD, where there is cumulative evidence for impaired contextualization as a key neurobiological underpinning. 5) Lack of geographical access to experts in exposure therapy, especially for PTSD, in rural areas.

DETAILED DESCRIPTION:
Anxiety and stress-related disorders are very common. One in three people experience some form of anxiety disorder including phobias, PTSD, and OCD. These disorders chronically limit one's ability to function and enjoy life. In addition to the common prevalence, wars in Iraq and Afghanistan have left about 13% of the returning veterans with combat PTSD, and even more with partial symptoms. Lifetime prevalence of PTSD is as high as 10% in women. Economic burden of anxiety disorders is between 42 to 52 billion dollars, one third of the country's total mental health bill. Near 30% of this money is spent in treatment costs. Burden of lost workdays only for PTSD is $3 billion. OCD affects 2.3% of the U.S. adults, half have serious impairment. Social phobia is one of the most common anxiety disorders with a 12 months prevalence of 6.8% and lifetime prevalence of 12.1%

Exposure therapy is the most effective treatment for cue-related anxiety disorders such as specific phobias, social phobia, OCD, and PTSD. The core principle is exposure to the feared objects/situations guided by a clinician. For example, in arachnophobia (fear of spiders) patient is exposed to picture of a spider on a computer, or from distance in the office, and gradually, with help of the clinician, they tolerate view of the spider from a closer distance. Clinician has a crucial role as the social safety cue in this process.

Although exposure therapy is very effective in treatment of phobias, OCD, and PTSD, there are limitations. Access and adherence to, and efficacy of exposure therapy are limited to 50% by multiple factors: First, there is a national shortage of psychiatrists and psychotherapists; patients often have to be on waiting list for weeks to months, and in many geographical locations such services are extremely scarce or do not exist. More than 50% of clinicians are not trained in exposure therapy, and there is usually geographical barriers for access to skilled therapists. In general, more than half of the US counties are unable to recruit mental health providers. Very frequently patients only receive medication or supportive therapy for several years before they can see a specialist trained in exposure therapy. Certain conditions like social phobia or PTSD make it increasingly difficult to leave the house and go to the clinic. Second, the feared objects are not always available in office for exposure and exposure most of the times is limited to pictures, movie clips, imagination, narrative, or memories. Imaginary exposure commonly lacks the level of arousal that is required for development of new safety learning. Third, patients have to practice real-life exposure on their own. In vivo treatment is commonly limited: often patients do not create situations that elicit the optimal safety learning, do not know how to create exposure situations, or simply do not follow through because of high anxiety in the absence of someone to coach them. This gap between exposure in the office, and real-life exposure remains a significant roadblock in successful exposure therapy. Fourth, clinicians are usually unable to provide treatment across multiple physical, temporal and social contexts that can promote contextualization of safety learning. Exposure mostly happens in the physical, emotional, social, and temporal context of the office visits. A fifth limitation is that current exposure therapy methods, do not address overgeneralization of the fear response.

Augmented Reality Augmented reality (AR) is the next wave of interactive human-computer technology that provides an opportunity of mixing virtually created objects with reality. Instead of creating a completely synthetic environment, AR adds virtually created objects to the real non-synthetic context. These elements become part of the real context, or cover some of its components. AR technology ultimately becomes less expensive than virtual reality (VR) technology because it does not require modeling the whole environment.

The investigators have developed a proof of concept prototype. The prototype that includes a scenario for treatment of fear of spiders (arachnophobia) and fear of snakes. Software platform connects the patient to a clinician who is located in the same or a different physical space, the patient wears the AR device, the clinician is able to see the patient's field of view, and positions a virtual spider/snake in the patient's environment, clinician determines direction/velocity of motions of the virtual spider/snake, clinician leads patient through the process of exposure therapy process until patient is desensitized to the view of the spider/snake. Exposure can then advance to higher number of spiders/snakes, or larger ones.

Subject Recruitment: Subject recruitment will happen at the Wayne State University (WSU) Department of Psychiatry and Behavioral Neurosciences (DPBN) psychiatry clinic, through flyers spread on the campus, and advertisement on Wayne State's student website. The investigators aim to pre-screen a minimum of 50 individuals. The actual number of participants to be enrolled is 50, and the investigators have a minimum pre-screening of 50 anticipating that some may not qualify.

Treatment will take place at the Stress, Trauma, and Anxiety Research Clinic at the WSU department of psychiatry in Detroit. Participants will do 1-4 sessions of augmented reality exposure therapy (ARET), each lasting 90 minutes. The first session will include a short refresher on principles of exposure therapy, and training the use of the AR equipment.

At any time the level of distress due to exposure is determined too high, both patient and the provider can abort the exposure. This will be done similarly to any other conventional exposure therapy method.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of specific phobia of animals (i.e. spiders or snakes), according to diagnostic and statistical manual version 5 (DSM-V) criteria. Both genders, ages 18-45, who are able and willing to consent for involvement in the study.

Exclusion Criteria:

* Subjects who refuse or are unable to consent to participate in the study.
* Active abuse of substances or meet criteria for substance use disorder in the past 6 months
* Current or previous diagnosis of psychotic disorder, schizophrenia, obsessive-compulsive disorder, bipolar disorder, mental retardation, active abuse of substances or meet criteria for substance use disorder in the past six months substance use, or PTSD.
* Unstable behavior that, in the opinion of the investigator, would place the subject at increased risk or preclude the subject's full compliance with or completion of the study, e.g. significant Axis II disorder or suicidal behavior.
* Visual or auditory disabilities limiting ability use of AR goggles
* Current use of antidepressant medications, mood stabilizers, or benzodiazepines
* History of seizures or a condition that would increase likelihood for seizures
* Serious medical or neurological illness
* Wards of the court

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arash Javanbakht, MD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State U Department of Psychiatry, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AR Therapy Intervention for Spider Phobia | No Treatment Control Group for Spider Phobia | AR Therapy Intervention for Snake Phobia | No Treatment Control Group for Snake Phobia
Started | 13 | 12 | 0 | 0
Completed | 13 | 12 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants with untreated arachnophobia (as determined by clinician interview) were recruited through flyers at medical clinics and online posts to a university forum. OF NOTE: No participants were recruited for snake phobia data collection due to the COVID-19 pandemic halting in-person research activities, therefore no data were collected for snake phobia.
Groups:
- AR Therapy Intervention for Spider Phobia; AR Therapy Intervention for Fear of Snakes: Augmented reality (AR) exposure therapy involves placing virtual objects in the participant's real environment as a method of exposure therapy. The AR therapy intervention group will complete an exposure therapy session using an augmented reality headset. The participant will work with the therapist, who will control the augmented reality paradigm and cater the exposure to the needs of the participant. The exposure therapy session will be as long as needed to reduce anxiety to low and stable levels, as measured by the participant's subjective units of distress.
- No Treatment Control Group for Spider Phobia; No Treatment Control Group for Fear of Snakes: This will be a waitlist control group that will receive no treatment for the duration of the study, however they will be offered the opportunity for some form of exposure therapy following the conclusion of the study (1 month).
- Total: Total of all reporting groups
Arm/Group | AR Therapy Intervention for Spider Phobia | No Treatment Control Group for Spider Phobia | AR Therapy Intervention for Fear of Snakes | No Treatment Control Group for Fear of Snakes | Total
Number analyzed (Participants) | 13 | 12 | 0 | 0 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 12 | 0 | 0 | 25
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 23 [18 to 45] | 24 [18 to 45] |  |  | 23.5 [18 to 45]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female | 9 | 7 | 0 | 0 | 16
  Sex: Male | 3 | 3 | 0 | 0 | 6
  Sex: Did Not Report | 1 | 2 | 0 | 0 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 12 | 0 | 0 | 25

OUTCOME MEASURES:

1. Primary Outcome: Spider Phobia
Description: Fear of spiders / severity of phobia will be measured via the Fear of Spiders questionnaire in order to determine how treatment has impacted the fear.
  The fear of spiders questionnaire is 18 items scored on a scale from 1-7, for a low score of 18 and a high score of 126. Total score is calculated by adding all items together. Higher scores are indicative of greater fear of spiders.
Time Frame: Change in score on Fear of Spiders questionnaire from baseline to post-treatment, at one month follow-up
Population: OF NOTE: No participants were recruited for snake phobia data collection due to the COVID-19 pandemic halting in-person research activities, therefore no data were collected for snake phobia.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AR Therapy Intervention for Spider Phobia | No Treatment Control Group for Spider Phobia | AR Therapy Intervention for Snake Phobia | No Treatment Control Group for Snake Phobia
Number analyzed (Participants) | 13 | 12 | 0 | 0
score on a scale
  Baseline Score | 104 (10.8) | 111 (11.7) |  |
  Post Treatment Score | 43.2 (22.5) | 102 (18.4) |  |
Statistical Analysis 1: Comparison: AR Therapy Intervention for Spider Phobia vs No Treatment Control Group for Spider Phobia; A repeated measures ANOVA was conducted to assess main effects of group (AR therapy intervention versus no treatment control), time (baseline, one week follow up, and one month follow up) as well as an interaction effect. The P-Value shown below is for the interaction effect. Post-hoc power analysis indicated actual power 99%, critical F=4.76; Test type: Superiority; p < .001, ANOVA — Interaction effect: p<.001, np2=.720; Main effect of time: p<.001, np2=.798; main effect of group: p<.001, np2=.711

2. Secondary Outcome: Behavioral Approach Test--Ability to Confront Phobia
Description: A measure of the closest distance the patient can have to the feared object. Scored from 0-12 based on distance away in meters from feared object and interaction with feared object. The score is given based on participant interaction, therefore one value is chosen. Higher values closer to 12 show greater comfortability and ability to interact with the feared object.
Time Frame: Change in score on Behavioral Approach Test from baseline to post-treatment, at one month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | AR Therapy Intervention for Spider Phobia | No Treatment Control Group for Spider Phobia | AR Therapy Intervention for Snake Phobia | No Treatment Control Group for Snake Phobia
Number analyzed (Participants) | 13 | 12 | 0 | 0
meters
  Baseline Distance | 6.27 (2.26) | 7.5 (5.16) |  |
  Post Treatment Distance | 0 (0) | 6 (3.03) |  |
Statistical Analysis 1: Comparison: AR Therapy Intervention for Spider Phobia vs No Treatment Control Group for Spider Phobia; A repeated measures ANOVA was conducted to assess main effects of group (AR therapy intervention versus no treatment control), time (baseline, one week follow up, and one month follow up) as well as an interaction effect. The P-Value shown below is for the interaction effect. Post-hoc power analysis indicated actual power 96%, critical F=4.76; Test type: Superiority; p < .001, ANOVA — Interaction effect: p<.001, np2=.542; Main effect of time: p<.001, np2=.598; and main effect of group: p<.001, np2=.439

3. Other Pre Specified Outcome: Snake Phobia
Description: Fear of snakes will be measured via the snake anxiety questionnaire. The Snake Anxiety questionnaire is a 30 item true or false questionnaire. The number of true or false responses are summed. Higher number of true responses is indicative of greater phobia.
Time Frame: Change in score on Snake Anxiety questionnaire from baseline to post treatment (immediately following the last exposure therapy session)
Population: as for outcome 1
Arm/Group | AR Therapy Intervention for Spider Phobia | No Treatment Control Group for Spider Phobia | AR Therapy Intervention for Snake Phobia | No Treatment Control Group for Snake Phobia
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Other Pre Specified Outcome: Spider Phobia--additional Measure
Description: The Spider Phobia questionnaire is a 31 item questionnaire with yes or no responses. All items are added together for a total score. 9 items are reverse scored. The minimum score is 0 and the maximum score is 31. Higher scores are indicative of more severe phobia. This questionnaire will serve as an additional measure of spider phobia to the primary outcome measure.
Time Frame: Change in score on Spider Phobia questionnaire from baseline to post-treatment, at one month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AR Therapy Intervention for Spider Phobia | No Treatment Control Group for Spider Phobia | AR Therapy Intervention for Snake Phobia | No Treatment Control Group for Snake Phobia
Number analyzed (Participants) | 13 | 12 | 0 | 0
score on a scale
  Baseline Score | 20.4 (4.25) | 25.7 (3.23) |  |
  Post Treatment Score | 11.1 (5.69) | 24.9 (3.14) |  |
Statistical Analysis 1: Comparison: AR Therapy Intervention for Spider Phobia vs No Treatment Control Group for Spider Phobia; A repeated measures ANOVA was conducted to assess main effects of group (AR therapy intervention versus no treatment control), time (baseline, one week follow up, and one month follow up) as well as an interaction effect. The P-Value shown below is for the interaction effect. Post-hoc power analysis indicated actual power 99%, critical F=3.49; Test type: Superiority; p < .005, ANOVA — Interaction effect: p<.005, np2=.481; Main effect of time: p<.001, np2=.572; and main effect of group p<.001, np2=.626

ADVERSE EVENTS:
Time Frame: Through study completion, approximately 1 month
Arm/Group | AR Therapy Intervention for Spider Phobia | No Treatment Control Group for Spider Phobia
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/47/NCT03649347/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/47/NCT03649347/SAP_001.pdf